CLINICAL TRIAL: NCT05444127
Title: Oral Health and Wilson's Disease: SOMAWI
Acronym: SOMAWI
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: APS_2022_5
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: patients with hepatic form of Wilson disease and those with neurological form
  Interventions: Other: Saliva samples; Other: Questionnaire OHIP-14; Other: Thorough dental examination
- controls: control population consulting in routine dental with panoramic dental imaging, outside of an emergency context
  Interventions: Other: Questionnaire OHIP-14; Other: Thorough dental examination

INTERVENTIONS:
Other: Saliva samples — A saliva sample is added by research for all patients, as well as an oral quality of life questionnaire. For the witnesses, participation also entails the completion of the standardized oral examination (potentially longer than the assessment that would have been carried out as part of the treatment) and the administration of the oral quality of life questionnaire.
  Groups: Cases
Other: Questionnaire OHIP-14 — A saliva sample is added by research for all patients, as well as an oral quality of life questionnaire. For the witnesses, participation also entails the completion of the standardized oral examination (potentially longer than the assessment that would have been carried out as part of the treatment) and the administration of the oral quality of life questionnaire.
Other: Thorough dental examination — A saliva sample is added by research for all patients, as well as an oral quality of life questionnaire. For the witnesses, participation also entails the completion of the standardized oral examination (potentially longer than the assessment that would have been carried out as part of the treatment) and the administration of the oral quality of life questionnaire.

SUMMARY:
Patients with Wilson disease have poorer dental and periodontal health and a have lower oral quality of life than control patients. Patients with a neurological form would also more frequently present limitations in the function of the masticatory apparatus. Systemic treatments for Wilson disease are associated with lesions of the oral mucosa. Analysis of copper level in saliva could testify to the effectiveness of copper depletion in treated patients The main objective is to compare the state of dental health between: patients with Wilson disease in the hepatic form and patients with the neurological form, and a population of controls.

DETAILED DESCRIPTION:
The comparaison between the three groups is based on evaluation criteria wich is CAOD index of caries severity (developed by Klein and Palmer in 1940) counting the number of permanent teeth with caries (evolving to include non-cavitary caries) (C), absent due to caries (A) and filled (O) in an individual. The maximum score is 28 (third molars are not taken into account). The index is obtained from clinical examination and panoramic dental imaging.

ELIGIBILITY:
Inclusion Criteria:

* Express consent to participate in the study
* Member of or beneficiary of a social security scheme
* For cases: Affected by Wilson's disease
* For controls: Benefiting from a first routine dental consultation with dental panoramic imaging, outside of an emergency context or treatment follow-up/maintenance

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding women
* Severe psychiatric disorders with behavioral disorders
* For cases:

  * hepatic or neurological decompensation
  * liver transplant patient
* For witnesses:

  * Patient with hepatic or neurological disease
  * Patient taking dietary supplements enriched with copper or zinc or zinc supplementation
  * Patient wearing removable prostheses with zinc-enriched prosthetic adhesives (Fixodent ProPlus®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruitment of Wilson patients will be done in the coordinating center of the CRMR Wilson at the Fondation A de Rothschild Hospital. Control patients matched in age and sex will be identified among patients consulting in the oral medicine department of Charles Foix Hospital. Posters will be placed in the waiting room to inform patients of the existence of the study and promote recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
CAOD index of the severity of the caries impairment counting the number of permanent teeth decayed in an individual. The maximum score is 28 (third molars are not taken into account) | inclusion visit
  The index is obtained from clinical examination and panoramic dental imaging

CONTACTS AND LOCATIONS:
Overall Officials: Marjolaine GOSSET, Study Director — Hopital Charles Foix
Locations (3):
- France (3):
  - Hopital Charles Foix, Ivry-sur-Seine
  - Hôpital Charles Foix, Ivry-sur-Seine
  - Fondation Adolphe de Rothschild, Paris